CLINICAL TRIAL: NCT01292889
Title: Gene Polymorphisms in Mood Disorders
Brief Title: Study of Genes in Relation to Seasonal Affective Disorder and Major Depressive Disorder
Acronym: Season605
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Kathryn Ariel Roecklein, Associate Professor, University of Pittsburgh
Other Study IDs: Seasonality605
Record Dates: First submitted 2011-02-08; First posted 2011-02-10 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Seasonal Affective Disorder
Keywords: Seasonal Affective Disorder; Major Depressive Disorder; Depression; Winter Blues
MeSH Terms: conditions — Seasonal Affective Disorder; Depressive Disorder, Major; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva samples for DNA collection
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Seasonal Affective Disorder: Consists of Individuals with Seasonal Affective Disorder
- Subsyndromal Seasonal Affective Disorder: Consists of individuals who do not meet SAD criteria,but present more symptoms for the disorder than do controls.
- Major Depressive Disorder: Consists of individuals who have MDD.
- Controls: Consists of individuals who do not present symptoms of SAD or MDD.

SUMMARY:
The investigators are looking for volunteers who have a history of Major Depressive Disorder, the Winter Blues, or Seasonal Affective Disorder or healthy volunteers who do not have a history of these disorders for a research study on genetics.

DETAILED DESCRIPTION:
The investigators are looking for volunteers who have a history of Major Depressive Disorder, the Winter Blues, or Seasonal Affective Disorder or healthy volunteers who do not have a history of these disorders for a research study on genetics. Participation involves one 2-3 hour visit involving two diagnostic interviews, DNA collection, and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* SAD or MDD
* healthy control

Exclusion Criteria:

* drug or alcohol dependence
* Bipolar Disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn A Roecklein, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Department of Psychology 605 Old Engineering Hall, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Summary data will be provided upon request to collaborators.